CLINICAL TRIAL: NCT03799523
Title: Demonstration of a Novel Approach Using Surface-Image Guidance to Improve Delivery of Breast Radiotherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CTMS# 18-0135; 18-769H (Other: UT Health Science Center Institutional Review Board)
Record Dates: First submitted 2018-11-19; First posted 2019-01-10 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subjects undergoing breast radiotherapy (Experimental): At the time of CT simulation study participants will receive temporary skin markings to be covered in clear medical grade tape. Light-based surface imaging will be used to determine alignment between the patient and the radiation machine. Radiation treatment will proceed as standard of care.
  Interventions: Other: Temporary skin markings; Other: Surface imaging

INTERVENTIONS:
Other: Temporary skin markings — To use temporary markings in lieu of localization tattoos.
Other: Surface imaging — To use light-based surface imaging for patient positioning during radiation treatment.

SUMMARY:
The first goal of this project is to validate the superiority of semi-permanent marks used in conjunction with specialized light-based surface imaging (SIGRT) in an effort to phase out the use of permanent tattoos for the investigator's patients. The secondary goal of this project is to validate the superiority of specialized light-based surface imaging for daily radiation set-up compared to standard-of-care imaging methods using ionizing radiation, such as weekly port films or cone-beam CT (CBCT) scans during a radiation therapy course for breast cancer.

DETAILED DESCRIPTION:
This study uses surface imaging for breast patients to standardize or normalize planning position & minimize variability of port films thus reducing systematic error. The primary objective of this study is to demonstrate the superiority of using surface imaging to combine an ideally gated treatment planning CT and verification images timed to the breathing cycle, quantified as the total within-subject variation of the measured location relative to current methods of radiation delivery not using this approach. The secondary objective is to demonstrate the superiority of specialized light-based surface imaging for daily radiation set-up without tattoos compared to standard-of-care methods with regard to the total within-subject variation of the measured location determined by weekly port films during a course of radiation for breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Biologically female
* Ability to provide informed written consent in either English or Spanish
* Surgical pathology and staging scans must demonstrate Ductal carcinoma in situ (DCIS) or invasive breast cancer, Stages 0, 1, 2, and 3
* Patient will undergo adjuvant radiation therapy as a part of multimodality breast cancer treatment with plans for tangent field radiation treatment with or without loco-regional lymph node targeting, based on the clinical judgement of the treating physician
* Willingness to maintain temporary skin markings for a part of their of radiation therapy duration
* Absence of any conditions that may affect ability to have either tattoos or skin markings, as discussed in Exclusion Criteria

Exclusion Criteria:

* Age < 18 years
* Biologically non-female
* Inability or unwillingness of subject to give written informed consent
* Patients found at presentation to have very locally-advanced cancer (e.g. inflammatory breast cancer) or metastatic breast cancer (Stage 4)
* Patients that will be treated with a deep-inspiration breath hold technique (typically younger patients being treated for left-sided tumors)
* Current pregnancy, as this is a contraindication to receiving radiation therapy
* History of prior radiotherapy to the chest wall or torso
* Known allergy / sensitivity to standard medical marking tattoo ink (by design non-toxic, low-allergy), skin marking paint, or medical tape (e.g. Tegaderm)
* Active drug or alcohol use or dependence evidenced by patient record and/or self-report that, in the opinion of the investigator, would interfere with adherence to daily radiation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Position measurement from Port films. | Once weekly for 3 weeks up to 5 weeks
  Distance measured (centimeters) from the planned position of radiotherapy to the actual position of radiotherapy on weekly port films. Port films are x-rays of the treatment field which are done to ensure that the patient and the radiation machine are properly aligned to each other. Weekly port films will be obtained for the duration of radiation treatment, which will be from three to five weeks in length.

CONTACTS AND LOCATIONS:
Overall Officials: Eva Galvan, MD, Principal Investigator — Principal Investigator
Locations (1):
- UT Health San Antonio Mays Cancer Center, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided